CLINICAL TRIAL: NCT04155476
Title: Ultrasound Evaluation of the Change in Diameter of the Posterior Tibial Artery and Dorsalis Pedis Artery After the Administration of Topical Nitroglycerin.
Brief Title: Ultrasound Evaluation of Lower Extremity Arteries After Topical Nitroglycerin Administration
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Deborah Heart and Lung Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2k19-09
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitroglycerin exposure (Experimental)
  Interventions: Drug: Nitroglycerin Topical Product
- Non-Nitroglycerin exposure (Placebo Comparator)
  Interventions: Drug: Nitroglycerin Topical Product

INTERVENTIONS:
Drug: Nitroglycerin Topical Product — application of NG topical to dorsals pedis and posterior tibial arteries.

SUMMARY:
There have not been any published studies showing the use of topical nitroglycerin on the dilatory effect on the posterior tibial or dorsalis pedis arteries. The objective of this study is to determine the response of the posterior tibial artery and dorsalis pedis artery to topical administration of nitroglycerin. This study may provide further information for the utility of this artery in the treatment of peripheral arterial disease.

DETAILED DESCRIPTION:
This will be a prospective, randomized, blinded, placebo-controlled study to gather data on the effect of nitroglycerin on the pedal artery of patients with varying comorbidities. Patients will be divided into a treatment group and a control group. A detailed history will be taken from the patient to ascertain risk factors such as Hypertension, Hyperlipidemia, CAD, PAD, Tobacco abuse, Diabetes Mellitus, Family history of CAD/PAD, or history of non-healing wounds. Further demographic data such as sex, age, height, weight, body surface area, and body mass index will be documented.

Ultrasound measurements of the dorsalis pedis and anterior tibial artery will be obtained at baseline. Measurements will be obtained in the perpendicular plane using B mode on the vascular ultrasound. The largest diameter will be documented. Measurement of the largest intima diameter will be obtainedThe image will be temporarily stored for measurement purposes but will not be saved. The patients will then have differing treatments based on their groupings into the control or treatments arms.

Patient history, demographics and artery measurements will be kept on a password protected document and assigned a research patient identifier number. Another password protected document will contain the patient's name and patient identifier number. Only the principal investigator and sub-principal investigators will have access to these documents.

Patients in the control group will have measurements of their posterior tibial artery or dorsalis pedis artery bilaterally. The sites of evaluation will be marked with a surgical marker. A topical moisturizer will be placed 1 cm proximal to the measured areas of the leg and covered with a dressing bilaterally. Measurements of the arteries will be made at baseline, 10 minutes, 30 minutes, 60 minutes, and 90 minutes. In addition, non-invasive Blood Pressure measurements will be made at baseline, 10 minutes, 30 minutes, 60 minutes, and 90 minutes. The Moisturizer will be removed at 60 minutes bilaterally.

Patients in the treatment group will again receive measurements of the posterior tibial and dorsalis pedis arteries bilaterally which will be marked with a surgical marker. Randomly, the tibial artery or dorsalis artery will be selected and nitroglycerin paste will be placed 1 cm proximal to the measured area of one leg and moisturizer will be placed on the other leg in order create uniformity. Both legs will be covered with a dressing. These patients will randomly receive 15mg or 30mg of nitroglycerin. Bilateral measurements of the posterior tibial and dorsalis pedis arteries will be made at baseline, 10 minutes, 30 minutes, and 60 minutes, 90 minutes. In addition, non-invasive Blood Pressure measurements will be made at baseline, 10 minutes, 30 minutes, 60 minutes, and 90 minutes in the arm. The Moisturizer and nitroglycerin will be removed at 60 minutes.

Data handling and record keeping:

All data collected, including demographic information will be kept in the Cardiology research department, in a cabinet with lock and key. All electronic documents will be password protected and encrypted. Only the principal investigator and sub-principal investigators will have access to data.

Quality control and quality assurance:

The posterior tibial artery will initially be localized utilizing palpation starting at the level of the medial malleolus. Positioning will subsequently be confirmed by the use of ultrasound.

The Dorsalis Pedis artery will be localized utilizing palpitation starting at the level of the navicular bone. Positioning will subsequently be confirmed by the use of ultrasound.

When possible there will be an attempt to use measurements at the level of the anatomical landmark in order to provide standardization Any deviation will be documented.

Assessment of the Posterior Tibial and Dorsalis pedis arteries diameter and administration of nitroglycerin.

A Vascular ultrasound probe will be used to evaluate the diameter of the arteries. The same vascular probe will be used to evaluate each patient to ensure standard measurements. A horizontal and vertical diameter will be obtained to obtain an "Averaged diameter". Subsequently, the level measured will be marked to ensure rapid and accurate re-evaluation of the same area.

Nitroglycerin paste or moisturizer will be added to the treatment/control leg/artery depending on the arm of the study the patient is randomized to. It will be administered 1 cm above the site being evaluated. Measurements will be made at 30, 60, and 90 minutes.

Risks:

Possible risks include hypotension (although this was not noted in prior studies using nitroglycerin in the radial artery), headache, rash, possible allergic reaction to any components.

Benefits:

The effects of nitroglycerin on dilatation and spasm of the radial artery has been previously documented. . As the pedal arteries become more widely used in the treatment of peripheral arterial disease, a quantification of the effects of nitroglycerin on the pedal arteries will be beneficial for its potential as an alternative or auxiliary access site in peripheral cases.

Safety:

This study is exclusively for inpatients. The half-life of nitroglycerin is 30 minutes. As a result, 2.5 hours after the ointment has been removed, the nitroglycerin will be considered metabolized. During this time the patient will be closely monitored. Only one patient will be investigated at a time and the investigator initiating the study will be present on the medical floor for the duration of the entire examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Deborah Heart & Lung Center.
* Patients 18 years of age and older.

Exclusion Criteria:

* Patients who do not have the ability to provide informed written consent.
* Patients with documented allergy to Nitroglycerin
* Recent/chronic use of nitrates/vasodilatory medications.
* Patients with a SBP <100, labile blood pressure, tachycardia, hemodynamic instability.
* Patients with recent admission requiring antibiotics.
* Patients who are pregnant or nursing.
* Patients who have current or chronic liver, renal, rheumatologic, or neurological disease. - Patients who have had peripheral vascular procedures in the prior 30 days.
* Patients who have had any procedure or operation during their current hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12-30 (Estimated); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Vessel Diameter after administration of NG topical | 3 months
  Determination of the diameter of the posterior tibial artery and dorsalis pedis artery before and after the administration of various doses of topical nitroglycerin.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Beyer AT, Ng R, Singh A, Zimmet J, Shunk K, Yeghiazarians Y, Ports TA, Boyle AJ. Topical nitroglycerin and lidocaine to dilate the radial artery prior to transradial cardiac catheterization: a randomized, placebo-controlled, double-blind clinical trial: the PRE-DILATE Study. Int J Cardiol. 2013 Oct 3;168(3):2575-8. doi: 10.1016/j.ijcard.2013.03.048. Epub 2013 Apr 10. PMID 23582415
- [Background] Majure DT, Hallaux M, Yeghiazarians Y, Boyle AJ. Topical nitroglycerin and lidocaine locally vasodilate the radial artery without affecting systemic blood pressure: a dose-finding phase I study. J Crit Care. 2012 Oct;27(5):532.e9-13. doi: 10.1016/j.jcrc.2012.04.019. Epub 2012 Jun 12. PMID 22699036
- [Background] Chong AY, Lo T, George S, Ratib K, Mamas M, Nolan J. The effect of pre-procedure sublingual nitroglycerin on radial artery diameter and Allen's test outcome - Relevance to transradial catheterization. Cardiovasc Revasc Med. 2018 Mar;19(2):163-167. doi: 10.1016/j.carrev.2017.07.016. Epub 2017 Jul 29. PMID 28923695